CLINICAL TRIAL: NCT04257149
Title: Mobile Microwave-based Diagnosis and Monitoring of Stroke: on the Road Towards Improved Stroke Triage and Care, Including Prehospital Initiation of Thrombolytic Treatment
Brief Title: Mobile Microwave-based Diagnosis and Monitoring of Stroke
Acronym: MODS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Haukeland University Hospital (Other); Equinor (Unknown); Medfield Diagnostics (Industry); Nordlandssykehuset HF (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SUSID663
Record Dates: First submitted 2018-02-01; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Stroke, Acute; Intracerebral Hemorrhage
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hemorrhagic stroke group (group A) (Experimental): Patient group A is defined as patients that are diagnosed with hemorrhagic stroke.
  Interventions: Diagnostic Test: Hemorrhagic stroke group (group A)
- Ischemic stroke group (group B) (Experimental): Patient group B is defined as patients that are diagnosed with ischemic stroke.
  Interventions: Diagnostic Test: Ischemic stroke group (group B)
- Stroke mimic group (group C) (Experimental): Patient group C is defined as patients with stroke mimics, i.e. with initially suspected stroke but not diagnosed with stroke.
  Interventions: Diagnostic Test: Stroke mimic group (group C)

INTERVENTIONS:
Diagnostic Test: Hemorrhagic stroke group (group A) — Group A: A microwave measurement (Stroke finder MD100) will be performed with the patient lying on the ambulance stretcher, in the hospital bed or another suitable surface.
  Arms: Hemorrhagic stroke group (group A)
Diagnostic Test: Ischemic stroke group (group B) — Group B: A microwave measurement (Stroke finder MD100) will be performed with the patient lying on the ambulance stretcher, in the hospital bed or another suitable surface.
  Arms: Ischemic stroke group (group B)
Diagnostic Test: Stroke mimic group (group C) — Group C: A microwave measurement (Stroke finder MD100) will be performed with the patient lying on the ambulance stretcher, in the hospital bed or another suitable surface.
  Arms: Stroke mimic group (group C)

SUMMARY:
This is a prospective, open, multicentre trial that will enrol patients with clinical signs of stroke in the acute phase admitted for CT scan. The study assesses the diagnostic capability and safety of Strokefinder MD100.

DETAILED DESCRIPTION:
This is a prospective, open, multicentre trial that will enrol patients with clinical signs of stroke in the acute phase admitted for CT scan. The investigator will assess and control the inclusion/exclusion criteria. If the patient is confirmed to be suitable for the trial, the patient is asked to give oral informed consent. If the answer is affirmative the microwave measurement will be performed. The procedure will take less than five minutes (the duration of the actual measurement procedure is 1.5 minutes) and will not interfere with the patient's standard of care during the hospital stay. Written informed consent is acquired by the investigator, as soon as possible after the acute phase of care is completed.

The measurement data will be evaluated for the presence of signal artifacts. The diagnostic ability of the device will be evaluated using a leave-one-out cross validation (LOOCV) method with the CT diagnosis as ground truth.

Safety will be evaluated throughout the trial, and a safety follow-up will be performed by the investigator 24 hours after the last microwave measurement. No further follow-up of patients is planned.

ELIGIBILITY:
Inclusion Criteria:

* Patient with clinical signs of stroke
* Patient should be ≥ 18 years of age
* Patient/next of kin confirms orally that the patient wants to participate in the trial (during acute phase)
* Signed Informed Consent Form (after acute phase)

Exclusion Criteria:

* Pregnant or nursing woman
* Fertile woman where pregnancy cannot be excluded
* Patient diagnosed with a condition associated with risk of poor protocol compliance
* The diagnostic procedure is deemed to interfere with the standard of care
* Any other condition or symptoms preventing the patient from entering the study, according to the investigator´s judgment
* Any patient that according to the Declaration of Helsinki is deemed unsuitable for study enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the diagnostic ability of the device to diagnose hemorrhagic stroke and ischemic stroke in the prehospital and hospital setting | Baseline
  The diagnostic ability as measured by the area under the curve of the device for patient groups (group C vs. groups A + B) using the LOOCV method

SECONDARY OUTCOMES:
Adverse events within 24 hours | Baseline to 24 hours
  Any adverse events occurring within 24 hours from the measurement procedure(s)
To evaluate the diagnostic ability of the device to differentiate patients with stroke mimics | Baseline
  To evaluate the diagnostic ability of the device to differentiate patients with stroke mimics from patients with stroke (hemorrhagic stroke and ischemic stroke) in the prehospital and hospital setting
To evaluate the delivery of adequate measurement data from the device | Baseline
  To evaluate the delivery of adequate measurement data from the device in the prehospital and hospital setting
To evaluate the amount of time needed to perform the measurement procedures | Basline
  To evaluate the amount of time needed to perform the measurement procedures in the prehospital and hospital settings

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kurz, PhD, Principal Investigator — Helse Stavanger HF
Locations (4):
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Norlandsykehuset HF, Bodø
  - Statoil As, Stavanger
  - Stavanger University Hospital, Stavanger

IPD SHARING:
Plan to Share IPD: No